CLINICAL TRIAL: NCT03669965
Title: A Two-Part, Randomized, Open-label, Multicenter, Phase 2a/2b Study of the Efficacy, Safety, and Pharmacokinetics of KRT-232 Compared to Ruxolitinib in Patients With Phlebotomy-Dependent Polycythemia Vera
Brief Title: KRT-232 Compared to Ruxolitinib in Patients With Phlebotomy-Dependent Polycythemia Vera
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-102
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A Arm 1 (Experimental): KRT-232 120mg by mouth once daily for Days 1-7, off treatment for Days 8-21 (21-day cycles)
  Interventions: Drug: KRT-232
- Part A Arm 2 (Experimental): KRT-232 240mg by mouth once daily for Days 1-7, off treatment for Days 8-21 (21-day cycles)
  Interventions: Drug: KRT-232
- Part A Arm 3 (Experimental): KRT-232 120mg by mouth once daily for Days 1-7, off treatment for Days 8-28 (28-day cycles)
  Interventions: Drug: KRT-232
- Part B KRT-232 Arm (Experimental): Recommended KRT-232 dose and schedule from Part A
  Interventions: Drug: KRT-232
- Part B Ruxolitinib Arm (Active Comparator): Ruxolitinib per approved prescribing label
  Interventions: Drug: Ruxolitinib
- Part A Arm 4b (Experimental): KRT-232 240mg by mouth once daily for Days 1-5, off treatment for Days 6-28 (28-day cycles)
  Interventions: Drug: KRT-232
- Part A Arm 2b (Experimental): KRT-232 240mg by mouth once daily for Days 1-7, off treatment for Days 8-28 (28-day cycles)
  Interventions: Drug: KRT-232

INTERVENTIONS:
Drug: KRT-232 — KRT-232, administered by mouth
  Arms: Part A Arm 1; Part A Arm 2; Part A Arm 2b; Part A Arm 3; Part A Arm 4b; Part B KRT-232 Arm
Drug: Ruxolitinib — Ruxolitinib per approved prescribing label
  Arms: Part B Ruxolitinib Arm

SUMMARY:
This study evaluates KRT-232, a novel oral small molecule inhibitor of MDM2, for the treatment of patients with phlebotomy-dependent polycythemia vera (PV). Inhibition of MDM2 in PV is a new mechanism of action in PV. In Part A, patients must be resistant or intolerant to hydroxyurea or have undergone treatment with interferon. In Part B, patients must be resistant or intolerant to hydroxyurea.

This study is a global, open-label Phase 2a/2b study to determine the efficacy and safety of KRT-232. In Part A of the study, patients will be randomly assigned to 5 arms with 2 different doses and 3 different dosing schedules of KRT 232. In Part B of the study, patients will be randomized either to treatment with KRT-232 administered at the recommended dose and schedule from Part A or to treatment with ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PV (WHO 2016)
* ECOG ≤ 2
* Part A: patients with and without splenomegaly are eligible
* Part A: patients must be resistant or intolerant to hydroxyurea or have undergone treatment with interferon
* Part B: only patients with splenomegaly are eligible
* Part B: patients must be resistant or intolerant to hydroxyurea

Exclusion Criteria:

* Diagnosis of post-PV myelofibrosis (IWG-MRT)
* Prior treatment with MDM2 inhibitors, p53-directed therapies, HDAC, BCL 2 inhibitors
* Splenic irradiation within 3 months prior to the first dose of study treatment
* Clinically significant thrombosis within 3 months of screening
* Grade 2 or higher QTc prolongation
* Part B: prior treatment with a JAK inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with splenomegaly achieving a response at Week 32 | 32 weeks
  Response defined as having achieved both of the following:
  * The absence of phlebotomy eligibility beginning at the Week 8 visit and continuing through Week 32, with no more than one phlebotomy eligibility occurring post-randomization and prior to the Week 8 visit
  * A reduction in spleen volume as assessed by MRI (or CT) ≥ 35% from baseline at Week 32

SECONDARY OUTCOMES:
Duration of response after achieving both the absence of phlebotomy eligibility and reduction in spleen volume (for patients with splenomegaly) | 4 years
Duration of response after achieving phlebotomy independence | 4 years
Change from baseline of MPN-SAF TSS v2.0 patient-reported outcome | 32 weeks
Change from baseline of EORTC-QLQ-C30 patient-reported outcome | 32 weeks

OTHER OUTCOMES:
Proportion of patients without splenomegaly achieving the absence of phlebotomy eligibility beginning at the Week 8 and continuing through Week 28, with no more than one phlebotomy eligibility occurring post-randomization and prior to Week 8 | 28 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Washington University School of Medicine, St Louis, Missouri
  - Gabrail Cancer Center, Canton, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
- Center Hospitalier Universitaire d'Angers, Angers, France
- Germany (4):
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Gemeinschaftspraxis Haematologie - Onkologie - Hauptstelle, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
- Békés Megyei Központi Kórház Pándy Kálmán Tagkórház, Gyula, Hungary
- Poland (2):
  - Dolnośląskie Centrum Transplantacji Komórkowych z Krajowym Bankiem Dawców Szpiku, Wroclaw, Lower Silesian Voivodeship
  - Szpital Wojewódzki w Opolu, Opole
- Spain (3):
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca